CLINICAL TRIAL: NCT00002341
Title: An Open-Label Extension Study of Maintenance Therapy in HIV-Positive Subjects With Fluconazole-Refractory Oropharyngeal Candidiasis Who Have Responded to Itraconazole Oral Solution
Brief Title: A Study of Treatments for Fungal Infections of the Mouth and Throat in HIV-Infected Patients Who Have Had Success With Itraconazole But Not With Fluconazole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 236C; ITR-USA-107
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Candidiasis, Oral; HIV Infections
Keywords: Itraconazole; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Candidiasis, Oral
MeSH Terms: conditions — Candidiasis, Oral; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
To provide maintenance treatment with itraconazole solution for patients who were clinical responders in the ITR-USA-94 protocol, even if they subsequently relapsed.

DETAILED DESCRIPTION:
Patients who responded to therapy on protocol FDA 236B receive maintenance with itraconazole oral solution for up to 6 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Met criteria for clinical response on protocol FDA 236B with no residual visible lesion of oropharyngeal candidiasis upon completion of that study OR had initial response on protocol FDA 236B with subsequent relapse and retreatment with itraconazole solution or other therapies.
* Life expectancy of at least 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Underlying clinical condition that would preclude completion of study or place subject at significant risk.
* Judged unreliable with respect to physician's directives.

Concurrent Medication:

Excluded:

* Rifampin.
* Rifabutin.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.
* Terfenadine.
* Astemizole.
* Systemic antifungals.

Patients with the following prior conditions are excluded:

* Previously documented disseminated candidiasis.
* Previous clinically significant adverse event during treatment with itraconazole oral solution, unless clearly attributable to an intercurrent illness or condition.
* History of significant hepatic abnormalities or clinical evidence of significant hepatic disease within 2 months prior to study entry.

Prior Medication:

Excluded:

* Any investigational drug (other than itraconazole solution) within 1 month prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Moskovitz B, Wu J, Baruch A, Benken C. Long term safety and efficacy of itraconazole oral solution (IS) for treatment of fluconazole refractory oropharyngeal candidiasis (OC) in HIV-positive patients (pts). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:124 (abstract no 325)
- [Background] Fessel WJ, Merrill KW, Ward D, Moskovitz B, Benken C, Oleka N, Grimwood H. Itraconazole oral solution (IS) for the treatment of fluconazole-refractory oropharyngeal candidiasis (OC) in HIV-positive patients. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:124 (abstract no 327)